CLINICAL TRIAL: NCT07304817
Title: Comparative Study on the Mode of Action of Vicadrostat and Spironolactone on Protein Profiles and Renal Hemodynamic Effects in Patients Chronic Kidney Disease With Cardiovascular Disease /Heart Failure
Brief Title: Comparative Study on the Mode of Action of Vicadrostat and Spironolactone on Protein Profiles and Renal Hemodynamic Effects (COMPARE-VS)
Acronym: COMPARE-VS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Boehringer Ingelheim (Industry); DELPHINIUM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COMPARE-VS; ECR COMPARE-VS (1378-0052) (Other Grant/Funding Number: Boehringer Ingelheim International GmbH); 2025-523743-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: CKD; Cardiovascular Diseases; Heart Failure
Keywords: COMPARE-VS; Spironolactone; Vicadrostat; CKD; mineralocorticoid receptor antagonist (MRA); aldosterone synthase inhibitor (ASi)
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — Spironolactone; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: A mechanistic trial using an open-label, parallel-group comparative design with 1:1 randomization and blinded endpoint assessment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicadrostat (Experimental): daily treatment with Vicadrostat and background Empagliflozin
  Interventions: Drug: vicadrostat / empagliflozin combination 1
- Spironolactone (Active Comparator): daily treatment with Spironlactone and background Empagliflozin
  Interventions: Drug: Spironolactone (drug)

INTERVENTIONS:
Drug: vicadrostat / empagliflozin combination 1 — Group 1
  Arms: Vicadrostat
Drug: Spironolactone (drug) — Group 2
  Arms: Spironolactone

SUMMARY:
In this study, investigators will compare the effect of vicadrostat combined with empagliflozin with the effect of spironolactone combined with empagliflozin on renal function and changes in protein profiles in blood and urine.

The hypothesis is that the renal and cardiac responses between vicadrostat and spironolactone differ due to mechanistic differences in their mode of action. Spironolactone is a mineralocorticoid receptor antagonist (MRA) and exerts its effect on a receptor, or a type of "receiver," found on various cells. Vicadrostat is an aldosterone synthase inhibitor (ASI) and inhibits aldosterone production. Therefore, both drugs affect aldosterone.

However, studies evaluating the differences between MRAs (such as spironolactone) and ASI (such as vicadrostat) and examining their effects on the kidneys in patients with chronic kidney disease with concurrent cardiovascular disease, and/or heart failure are still lacking.

For this study, all participants will be divided into two groups:

* Group 1. Participants in this group will receive one tablet of vicadrostat (10 mg) and one tablet of empagliflozin (10 mg) daily for 26 weeks.
* Group 2. Participants in this group will receive one tablet of spironolactone (25 mg) and one tablet of empagliflozin (10 mg) daily for the first four weeks. Participants in this group will then receive two tablets of spironolactone (50 mg) and one tablet of empagliflozin (10 mg) daily for the remaining 22 weeks. The spironolactone dosage may be adjusted during the study period (from 12.5 to 50 mg) based on blood test results.

DETAILED DESCRIPTION:
The hypothesis is that renal and cardiac response to a mineralocorticoid receptor antagonist (MRA) differs from the response to an aldosterone synthase inhibitor (ASi) due to the mechanistic differences in action between these two compounds. However, direct head-to-head comparative studies evaluating the renal, cardiac, and systemic effects of MRAs and ASi in patients with chronic kidney disease (CKD), with concomitant cardiovascular disease (CVD) or heart failure (HF), are lacking.

The main objective of this study in patients with chronic kidney disease with either cardiovascular disease and/or or heart failure is to compare the effects of the ASi, vicadrostat, with the steroidal MRA, spironolactone, on the change in kidney function from baseline to 4 and 26 weeks.

Secondary objectives include

* Change in renal hemodynamic measurements from baseline to 4 and 26 weeks
* Changes in plasma and urinary protein profiles and associated pathways from baseline to 4 and 26 weeks

This is a mechanistic trial using an open-label, parallel-group comparative design with 1:1 randomization and blinded endpoint assessment.

Treatment with vicadrostat (Investigational Medicinal Product; IMP 10mg daily) or spironolactone (Comparator IMP; 25-50mg daily) for 26 weeks whilst on empagliflozin (Auxiliary Medicinal Product; AxMP 10mg daily). In half of the enrolled subjects (targeted 50 subjects) renal hemodynamic measurements will be performed at baseline, at 4 and at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written and dated informed consent for participation prior to trial admission,
2. Age ≥18 years, female or male
3. Patients with

   * Heart failure*1 (any LVEF) and eGFR*2 between 25-90 mL/min/1.73m2 OR
   * Established cardiovascular disease*3 and eGFR between 25-60 mL/min/1.73m2 OR
   * Established cardiovascular disease and type 2 diabetes and eGFR between 25-90 mL/min/1.73m2
4. Serum potassium ≤ 5.0 mmol
5. Currently treated or eligible for treatment with Empagliflozin*4
6. Not using a MRA or AS inhibitor in the last 6 months prior to enrollment
7. On stable doses of other guideline directed medical therapies for ≥ 4 weeks prior to enroll-ment
8. Outpatient.

   * 1 HF is defined as the definition used in the most recent ESC guidelines for HF.
   * 2 eGFR as assessed by the 2009 CKD-EPI without the race coefficient
   * 3 Cardiovascular disease is defined as a history of a myocardial infarction, coronary bypass surgery, PCI, or proven coronary artery disease (e.g. by coronary angiography, CT-scan, etc.)
   * 4 If switching from another SGLT2i to Empagliflozin subjects can be enrolled directly. If the subject is not yet on SGLT2i and starts Empagliflozin enrollment can start 4 weeks later see criteria 8.

Exclusion Criteria:

1. Inability to understand and sign informed consent
2. Absolute contra-indication for aldosterone antagonist
3. Absolute contra-indication for a SGLT2-inhibitor
4. Heart failure hospitalization, acute coronary syndrome, cardiac surgery, stroke or transient is-chemic attack in the 90 days prior to enrollment
5. Women who are pregnant, breastfeeding or may be considering pregnancy during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Kidney function (eGFR) | From baseline to 4 and 26 weeks of treatment.
  Changes in kidney function as determined by change in eGFR

SECONDARY OUTCOMES:
Renal hemodynamic measurements | From baseline to 4 and 26 weeks of treatment
  Changes in renal hemodynamic measurements
Plasma protein profiles | From baseline to 4 and 26 weeks of treatment
  Plasma protein profiles via proteomics
Urinary protein profiles | From baseline to 4 and 26 weeks of treatment
  Urinary protein profiles via proteomics
Changes in blood concentration markers | From baseline to 4 and 26 weeks of treatment
  Changes in blood (serum and plasma) concentrations of potassium, creatinine, neutrophil gelatinase-associated lipocalin (NGAL), renin, angiotensin II, aldosterone, and kidney injury molecule-1 (KIM-1).
Changes in urinary concentration markers | From baseline to 4 and 26 weeks of treatment
  Changes in urinary concentration of sodium, neutrophil gelatinase-associated lipocalin (NGAL), and kidney injury molecule-1 (KIM-1)
Changes in UACR | From baseline to 4 and 26 weeks.
  Changes in UACR

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Delphinium, Groningen, Provincie Groningen
  - University Medical Center Groningen, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided
will be updated at a later stage